CLINICAL TRIAL: NCT00183924
Title: A Phase II Pilot Study of Estramustine, Docetaxel, and Carboplatin for Patients With Hormone Refractory Prostate Cancer Progressing After Mitoxantrone-Based Chemotherapy.
Brief Title: Estramustine, Docetaxel, and Carboplatin for Patients With Hormone Refractory Prostate Cancer Progressing After Mitoxantrone-Based Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-01-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Estramustine; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Estramustine
Drug: Docetaxel
Drug: Carboplatin

SUMMARY:
This study is for patients with prostate cancer that is metastatic, progressive, and resistant to hormonal manipulation and mitoxantrone chemotherapy.Patients have previously been treated with surgical removal of the testes or hormone therapy, and subsequently with chemotherapy that included the drug, mitoxantrone (Novantrone). Patients will have prostate cancer that has worsened despite these treatments.

We hope to learn whether the combination chemotherapy decreases cancer symptoms and tests, and to determine how frequently serious side effects occur with acceptable toxicity from the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have had a histological diagnosis of adenocarcinoma of prostate and currently must have metastatic disease (stage TxNxM1) that is unresponsive or refractory to hormone therapy and mitoxantrone-based chemotherapeutic regimens. Patients must have metastatic prostate cancer deemed to be hormone- and mitoxantrone refractory by one or more of the following (despite androgen ablation, anti-androgen withdrawal and mitoxantrone therapy where applicable):

  1. Progression of measurable disease assessed within 28 days prior to registration.
  2. Progression of non-measurable (i.e. bone scan or PET scan) disease assessed within 42 days prior to registration.
  3. Rising PSA - defined as at least 2 consecutive rises in PSA documented over a reference value (measure 1). The first rising PSA (measure 2) should be taken at least 7 days after the reference value. A third confirmatory PSA measure is required (2nd beyond the reference level) to be greater then the second measure and it must be obtained at least 7 days after the 2nd measure. Patient must have a PSA concentration of at least 10 ng/ml in addition to increasing PSA to be eligible based on PSA criteria alone. No minimum PSA is required for patients with measurable disease or non-PSA evaluable disease.
* Age > 18 years
* Must have pre-study PSA (within 28 days prior to registration) Note: The PSA result (done within 28 days prior to registration) need not be elevated for inclusion provided other criteria for progression are met.
* Must have received prior hormonal therapy and have a castrate level of testosterone. Patients treated with orchiectomy are eligible. If they have been treated with non-steroidal anti-androgens, the patients must have ceased taking flutamide or nilutamide at least 28 days prior to enrollment and at least 42 days prior to enrollment for bicalutamide, and patients must have demonstrated disease progression. Either method of castration can have been supplemented with nonsteroidal antiandrogen (e.g. flutamide, bicalutamide, nilutamide).
* Must have received prior mitoxantrone therapy
* Prior radiation therapy is allowed but it must have been to less than 25% of total body bone marrow (see Appendix 5). This includes prior use of samarium, but patients cannot have received strontium. (>28 days must have elapsed since completion of RT with recovery from side effects. Soft tissue disease irradiated in the prior 2 months is not and may not be designated as measurable disease).
* May have received prior surgery (21 days must have elapsed since completion of surgery with recovery from side effects)
* Creatinine less than or equal to 1.5x the institutional upper limit of normal (within 28 days prior to registration)
* Bilirubin less than or equal to the institutional upper limit of normal (within 28 days prior to registration).
* Liver enzymes: If alkaline phosphatase is less than or equal to 4 x institutional upper limit of normal (ULN), then AST and ALT must be less than or equal to 2.0 x ULN. If alkaline phosphatase is > 4 x ULN in patients with bone metastases, then AST and ALT must be < 1.25 x ULN.
* Adequate bone marrow function. Complete blood count with differential must be done within 14 days prior to registration

  1. WBC greater than or equal to 3000 cells/mm3
  2. Absolute neutrophil count greater than or equal to 1500 cells/mm3
  3. Platelet count greater than than or equal to 100,000 cells/mm3
  4. Hemoglobin greater than or equal to 9.0 g/dl
* ECOG performance status 0-3. (For patients with PS of 3, cause must be due to pain secondary to bone metastases to be eligible)
* Must have pain (or be controlled on treatment for pain) attributable to metastatic prostate cancer as defined by a PPI score greater than or equal to 1. Subjects must have stabilization of their analgesic medications for at least one week prior to receiving study medication.
* No other chemotherapy, biological response modifiers, RT, radioisotope therapy (e.g. samarium or strontium), corticosteroid (>10mg of prednisone per day or equivalent), bisphosphonates or concomitant hormonal therapy may be given during protocol treatment. Patients may be treated with bisphosphonates provided they are initiated prior to study entry.
* Completed baseline QOL measures prior to registration (EORTC QLQ-C30 plus prostate cancer module; McGill Pain Questionnaire; Pain Medication Log. The nurse or CRA must complete QOL Cover sheet for baseline assessment prior to registration. Patient must be willing to complete other questionnaires while on study. If unable to complete questionnaires in English or Spanish, patient can be registered without contributing to QOL study).
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period (90 days) thereafter.
* Patients must be available for treatment and follow-up of any objective responses and/or residual toxicities.
* Willing and able to give informed consent and have signed an IRB approved informed consent

Exclusion Criteria:

* Myocardial infarction or angina pectoris within one year of registration
* History of brain metastases or currently has treated or untreated brain metastasis. (Patients with neurological symptoms must have CT or MRI brain negative for metastatic disease within 56 days prior to registration)
* Active thrombophlebitis or hypercoagulability.
* Known history of pulmonary embolism or deep venous thrombosis.
* Not recovered from major infections and/or surgical procedures, or has significant active concurrent other medical illness precluding protocol therapy or survival.
* Known or anticipated severe hypersensitivity reaction to estramustine, docetaxel, polysorbate 80 or carboplatin
* Other prior malignancy (except patients who have had another stage I or II malignancy currently in complete remission or other cancer with no evidence of disease for greater than 5 years from accrual to the current trial. Patients with basal or squamous cell carcinoma of the skin that have been treated with curative intent can be accrued to this trial 30 days after treatment).
* Preexistent peripheral neuropathy greater than or equal to grade 2
* Prior therapy with estramustine, taxanes (e.g. paclitaxel, docetaxel) or platinum-based (e.g. cisplatin, carboplatin, oxaliplatin) drugs or ongoing therapy
* Ongoing therapy with drugs known to inhibit P4503A4 drug metabolism including: Macrolide antibiotics: erythromycin, troleandomycin, azithromycin; Calcium antagonists: nifedipine, diltiazem; Imidazole antifungal agents: ketoconazole, itraconazole, fluconazole; HIV protease inhibitors; Immunosuppressive agents: cyclosporin, FK-506
* Ongoing therapy with drugs known to induce P4503A4 drug metabolism including: Phenobarbital, phenytoin, carbamazepine, griseofuvin and rifampin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-03; Primary Completion 2006-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Quinn, MD, Principal Investigator — University of Southern California
Locations (1):
- Norris Comprehensive Cancer Center, Los Angeles, California, United States